CLINICAL TRIAL: NCT01562561
Title: Multi-centre, Multinational, Open-labelled, Randomised, Parallel, Controlled Trial in Type 2 Diabetic Subjects Inadequately Controlled on Repaglinide, to Compare the Efficacy and Safety of Repaglinide Combined With Bedtime NPH Insulin Versus Twice Daily NPH Insulin
Brief Title: Efficacy and Safety of Repaglinide Combined With Insulin NPH in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGEE-1272
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rep + NPH (Experimental)
  Interventions: Drug: repaglinide; Drug: insulin NPH
- NPH (Active Comparator)
  Interventions: Drug: insulin NPH

INTERVENTIONS:
Drug: repaglinide — 2 mg at each main meal
  Arms: Rep + NPH
Drug: insulin NPH — Administrated subcutaneously (s.c., under the skin) either at bedtime or twice daily at breakfast and before dinner.

SUMMARY:
This trial is conducted in Asia and South Africa. The aim of this trial is to compare the efficacy and safety of repaglinide plus insulin NPH (insulin Neutral Protamine Hagedorn) with insulin NPH alone in subjects with type 2 diabetes inadequately controlled on repaglinide.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* HbA1c (glycosylated haemoglobin): 7-13% (both inclusive)
* BMI (body mass index) maximum 35 kg/m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2001-06-01 (Actual); Primary Completion 2002-12-20 (Actual); Study Completion 2002-12-20 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin) | Week 0 (visit 5); week 26

SECONDARY OUTCOMES:
FPG (fasting plasma glucose) | Week 0 (visit 5); week 26
7-point blood glucose profile | Week 0 (visit 5); week 26
Hypoglycaemic episodes | Week 0 (visit 5); week 26
Adverse events | Week 0 (Visit 5); week 26

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (12):
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Novo Nordisk Investigational Site, Kota Bharu, Kelantan, Malaysia
- Philippines (3):
  - Novo Nordisk Investigational Site, Marikina City
  - Novo Nordisk Investigational Site, Pasig
  - Novo Nordisk Investigational Site, Quezon City
- South Africa (6):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Alberton
- Novo Nordisk Investigational Site, Tainan, Taiwan

REFERENCES:
- [Result] Panelo A, Wing JR; AGEE-1272 Study Group. Repaglinide/bedtime NPH insulin is comparable to twice-daily NPH insulin. Diabetes Care. 2005 Jul;28(7):1789-90. doi: 10.2337/diacare.28.7.1789. No abstract available. PMID 15983336
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com